CLINICAL TRIAL: NCT04405986
Title: Exploring Brain Damages After COVID-19 Infection
Acronym: BRAINCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2020/20
Record Dates: First submitted 2020-05-08; First posted 2020-05-28 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV 2
Keywords: COVID-19; Brainstem; Electrophysiology
MeSH Terms: conditions — COVID-19 | interventions — Evoked Potentials, Auditory; Blinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrophysiological procedure (Experimental): Brainstem reflexes and neural conduction will be explored using Auditory Evoked Potentials (AEP) and blink and Masseter Inhibitory Reflex (MIR) in hospitalised patients with COVID infection
  Interventions: Procedure: Auditory Evoked Potentials (AEP); Procedure: Blink and Masseter Inhibitory Reflex

INTERVENTIONS:
Procedure: Auditory Evoked Potentials (AEP) — Record of electrophysiological responses (Auditory Evoked Potentials or AEP) during auditory stimulations with an electroencephalogram (EEG).
Procedure: Blink and Masseter Inhibitory Reflex — Electrophysiological exploration while stimulating trigeminal nerve to record 1) motor response induced (muscle contraction delay (Blink)) of the facial nerve, or 2) the contraction inhibition of masseters (Masseter Inhibitory Reflex (MIR)).

SUMMARY:
Although direct evidence is currently lacking, the high identity between SARS-CoV-1 and SARS-CoV-2 suggests, that the latter viral strain could also infect the Central Nervous System (CNS). Indeed, some cases of SARS-COV2 encephalitis begin to be described and CNS damages are increasingly highlighted in the literature, but still not objectified by imaging and do not allow to explain the entire clinical patterns. We hypothesise that these CNS damages are not always objectified by Magnetic Resonance Imaging (MRI) but could be indirectly observed by a physiological dysfunction of neural conduction in the brainstem. We will explore brainstem disruption through an electrophysiological approach.

DETAILED DESCRIPTION:
Clinical and preclinical data from studies with other coronaviruses suggest an evident neurotropism, which may result in more complex clinical scenarios. Can the SARS-CoV-2 enter the Central Nervous System (CNS) and infect neural cells ? And if yes, how the CNS damage contributes to pathophysiology of the COVID-19, to its signs, symptoms and progression as well as to its sequelae. It has been demonstrated that coronaviruses such as SARS-CoV and MERS-CoV do not limit their presence to the respiratory tract and frequently invade the CNS. The intranasal administration of SARS-CoV-1 or MERS-COV resulted in the rapid invasion of viral particles into the brain of mice, possibly through the olfactory bulb via trans-synaptic route. The brainstem, which hosts the respiratory neuronal circuit in the medulla, was severely infected with both types of viruses, which may contribute to degradation and failure of respiratory centres.

ELIGIBILITY:
Inclusion Criteria :

* Age ≥ 18 years.
* Hospitalized patient suffering from a positive COVID 19 diagnosed by Reverse transcription polymerase chain reaction (RT-PCR) or chest computed tomography scan (CTscan) with specific lesions

Exclusion Criteria :

* History of neurological damage interfering with auditory evoked potentials (PEA) and Electromyography (EMG) reflexes of the brainstem (stroke of the brainstem, acoustic neuroma, amyotrophic lateral sclerosis, facial diplegia, damage to nerves V or VII, etc.)
* Impaired alertness
* Sedative treatments or treatments that disturb nerve conduction.
* Pregnancy or breastfeeding
* Individuals under legal protection or unable to express personally their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Latency of electrophysiological response | Inclusion (T0)
  Latencies of electrophysiological responses with Auditory Evoked Potentials
Delay of Muscle contraction | Inclusion (T0)
  Delay of Muscle contraction (Blink reflex)
Delay of silent period | Inclusion (T0)
  Delay of silent period while the patient is asked to tighten the jaws (Masseter Inhibitory Reflex)
Duration of silent period | Inclusion (T0)
  Duration of silent period while the patient is asked to tighten the jaws (Masseter Inhibitory Reflex)
Inhibition rate | Inclusion (T0)
  Inhibition rate while the patient is asked to tighten the jaws (Masseter Inhibitory Reflex)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Glize, Principal Investigator — bertrand.glize@chu-bordeaux.fr
Locations (1):
- CHU de Bordeaux, Bordeaux, France